CLINICAL TRIAL: NCT03467542
Title: PHIL dAVF: Study of PHIL® Embolic System In The Treatment of Intracranial Dural Arteriovenous Fistulas
Brief Title: PHIL in the Treatment of Intracranial dAVF.
Acronym: PHIL dAVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL11005
Record Dates: First submitted 2018-03-06; First posted 2018-03-16 (Actual); Results first posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-05

CONDITIONS: Arteriovenous Dural Fistula
Keywords: Fistula; Intracranial; Dural; Arteriovenous; Liquid Embolic
MeSH Terms: conditions — Central Nervous System Vascular Malformations; Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- dAVF treatment (Experimental): PHIL® Liquid Embolic System
  Interventions: Device: PHIL® Liquid Embolic System

INTERVENTIONS:
Device: PHIL® Liquid Embolic System — The PHIL Embolic System is indicated in the treatment of dural arteriovenous fistulas (DAVF)

SUMMARY:
This study is a prospective, multicenter, single-arm study. Patients with Dural Arteriovenous Fistulas (dAVF) have a few choice for safe treatment. In this study, all patients with qualifying dAVFs will be treated with PHIL® Liquid Embolic material.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 - 80 years.
* Subject is willing and capable of complying with all study protocol requirements, including specified follow-up period.
* Subject or authorized legal representative must provide written informed consent prior to initiation of any study procedures.
* Subject has an intracranial dAVF

Exclusion Criteria:

* Subject having multiple dAVFs to be treated.
* Subject with a history of life threatening allergy to contrast media (unless treatment for allergy is tolerated).
* Subject has known allergies to dimethylsulfoxide, iodine.
* Subject is currently participating in another clinical study
* Female subject is currently pregnant.
* Subject has co-morbid conditions that may limit survival to less than 24 months.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, Principal Investigator — Mt. Sinai; Alan Boulos, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | dAVF Treatment
Started | 62
Completed | 60
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | dAVF Treatment
Number analyzed (Participants) | 62
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 56.6 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 45
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Neurological Death or Ipsilateral Stroke
Description: Reported incidences of death or ipsilateral stroke
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | dAVF Treatment
Number analyzed (Participants) | 62
Participants | 0
Statistical Analysis 1: Comparison: dAVF Treatment; Test type: Other; The total number evaluated, the percent, and the Clopper-Pearson two-sided 95% confidence limits on the percent

2. Secondary Outcome: Technical Events During the PHIL Embolization Procedure(s)
Description: Reported incidences of technical events with PHIL device
Time Frame: During the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | dAVF Treatment
Number analyzed (Participants) | 62
Participants | 0

3. Secondary Outcome: Device-related Adverse Events
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | dAVF Treatment
Number analyzed (Participants) | 62
Participants | 1

ADVERSE EVENTS:
Time Frame: 6 months after last embolization
Arm/Group | dAVF Treatment
All-Cause Mortality (participants affected / at risk) | 1/62
Serious Adverse Events (participants affected / at risk) | 5/62
Other Adverse Events (participants affected / at risk) | 27/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | dAVF Treatment (N=62)
Acute myocardial infarction (Cardiac disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Aortic dissection (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | dAVF Treatment (N=62)
dysacusis (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Diplopia (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Swelling face (General disorders) | 1
Ear infection (Infections and infestations) | 1
Radiation alopecia (Injury, poisoning and procedural complications) | 4
Procedural nausea (Injury, poisoning and procedural complications) | 2
Vascular site access hematoma (Injury, poisoning and procedural complications) | 1
Urinary retention post operative (Injury, poisoning and procedural complications) | 1
Vascular access site pseudo aneurysm (Injury, poisoning and procedural complications) | 1
Urinary tract procedural complication (Injury, poisoning and procedural complications) | 1
Vascular access site pain (Injury, poisoning and procedural complications) | 1
Procedural headache (Injury, poisoning and procedural complications) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 6
Procedural headache (Nervous system disorders) | 3
Seizure (Nervous system disorders) | 2
Transient Ischemic Attack (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Ischemic stroke (Nervous system disorders) | 1
Cerebral vasoconstriction (Nervous system disorders) | 1
Facial paresis (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Papillo edema (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator may publish the results if Sponsor has not published within eighteen (18) months after FDA approval of the Trial Devices.

The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03467542/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT03467542/SAP_001.pdf